CLINICAL TRIAL: NCT05686226
Title: A Phase II Trial of T Cell Receptor Gene Therapy Targeting Human Papillomavirus ( HPV) 16 E7 for HPV-Associated Cancers
Brief Title: E7 TCR-T Cell Immunotherapy for Human Papillomavirus (HPV) Associated Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Hinrichs (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Christian Hinrichs, Chief, Section of Cancer Immunotherapy, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192204; U01CA287904 (NIH); NCI-2023-02813 (Registry Identifier: [Registry ID: CTRP (Clinical Trial Reporting Program)]); Pro2022002259 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-12-25; First posted 2023-01-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Throat Cancer; Oropharynx Cancer; Anal Cancer; Vulva Cancer; Vaginal Cancer; Penile Cancer; Metastatic Cancer; HPV-Related Malignancy; HPV-Related Carcinoma; HPV-Related Cervical Carcinoma; HPV-Related Squamous Cell Carcinoma; HPV-Related Adenocarcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma; HPV-Associated Vaginal Adenocarcinoma; HPV-Related Adenosquamous Carcinoma; HPV-Related Endocervical Adenocarcinoma; HPV-Related Anal Squamous Cell Carcinoma; HPV-Related Penile Squamous Cell Carcinoma; HPV-Related Vulvar Squamous Cell Carcinoma; HPV Positive Rectal Squamous Cell Carcinoma
Keywords: Chimeric antigen receptors (CAR-T); Tumor infiltrating lymphocyte; TCR-T; immunotherapy; T cell; adoptive cell therapy; cellular therapy; gene therapy; human papillomavirus; HPV; E7; T cell receptor; TCR; E7 TCR; lymphocyte; cell therapy; cervical cancer; oropharyngeal cancer; anal cancer; vulvar cancer; vaginal cancer; penile cancer; tumor infiltrating lymphocytes (TIL); TIL therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Anus Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Penile Neoplasms; Neoplasm Metastasis | interventions — Adoptive Transfer; aldesleukin

STUDY DESIGN:
Intervention Model Description: This is a single-arm phase II clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- E7 TCR-T cells (Experimental): Subjects will receive a conditioning regimen, E7 TCR-T cells, and aldesleukin.
  Interventions: Biological: E7 TCR-T cells; Drug: Aldesleukin

INTERVENTIONS:
Biological: E7 TCR-T cells — Participants will receive a conditioning regimen consisting of cyclophosphamide and fludarabine. E7 TCR-T cells will be administered as a single intravenous infusion.
  Other Names: E7 TCR; HPV TCR; TIL; Adoptive cell transfer; CAR-T; TCR
Drug: Aldesleukin — Within 24 hours after E7 TCR-T cell infusion, aldesleukin 720,000 IU/kg IV every eight hours will be administered for up to six doses. Aldesleukin dosing will be stopped for aldesleukin-related grade 3 or greater toxicity other than flushing, fever, chills, or hemodynamic changes (tachycardia or hypotension) that respond to crystalloid infusion. Aldesleukin may also be stopped at any time at investigator discretion.
  Other Names: Proleukin

SUMMARY:
This is a phase II clinical trial to assess the clinical activity of immunotherapy with E7 TCR-T cells for metastatic HPV-associated cancers. HPV-associated cancers in include cervical, throat, penile, vulvar, vaginal, anal, and other cancers. Participants will receive a conditioning regimen, E7 TCR-T cells, and aldesleukin. Clinical response to treatment will be determined.

DETAILED DESCRIPTION:
This study will determine the tumor response rate for the treatment of HPV-associated cancers with E7 TCR-T cells. E7 TCR-T cells are autologous gene-engineered T cells that target HPV16 E7 through a T cell receptor (TCR). E7 is an HPV oncoprotein that is present in HPV-associated cancers. Participants must have the HLA-A*02:01 allele, which is required for tumor targeting by the E7 TCR. Treatment consists of a conditioning regimen (cyclophosphamide and fludarabine), a single infusion of E7 TCR-T cells, and adjuvant aldesleukin. Tumor response rate and response duration will be determined. Safety data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or refractory/recurrent HPV-16+ cancer.
2. Tumor with HPV16 genotype as determined by testing performed in a CLIA certified laboratory.
3. HLA-A*02:01 allele as determined by testing performed in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory. Participants may be enrolled based on low resolution typing (i.e., HLA-A*02) but the HLA-A*02:01 allele type must be confirmed prior to apheresis.
4. Measurable disease as assessed by RECIST Criteria Version 1.1.
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at screening.
7. Must have received prior first line standard therapy or have declined standard therapy.
8. Standard treatment options for first and second-line therapy must be presented and formally declined (Appendix VII).
9. Patients with three or fewer brain metastases that have been treated with surgery or stereotactic radiosurgery are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month before protocol treatment. Patients must be fully recovered from surgery.
10. Negative pregnancy test for women under 55 and all women who have had a menstrual period in the last 12 months. A pregnancy tests is not required for women who have had a bilateral oophorectomy or hysterectomy.
11. Men and women of child-bearing potential must agree to use adequate contraception (i.e., intrauterine device, hormonal barrier method of birth control; abstinence; tubal ligation or vasectomy) prior to study entry and for four months after treatment. Should a women become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
12. Seronegative for HIV antibody, hepatitis B antigen, and hepatitis C antibody. If a hepatitis C antibody test is positive, then testing for antigen by RT-PCR for Hepatitis C (HCV) RNA must be negative.
13. Participants must have organ and marrow function as defined below:

    1. Leukocytes > 3,000/microliter (mcL)
    2. Absolute neutrophil count > 1,500/mcL
    3. Platelets > 100,000/mcL
    4. Hemoglobin > 9.0 g/dL
    5. Total bilirubin within normal institutional limits except in participants with Gilbert's Syndrome who must have a total bilirubin < 3.0 mg/dL.
    6. Serum aspartate transferase (AST) (SGOT)/alanine transaminase (ALT) (SGPT) < 2.5 x upper limit of normal (ULN)
    7. Calculated creatinine clearance (CrCl) >50 mL/min/1.73 m2for participants with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation).
    8. international normalized ratio (INR) or activated partial thromboplastin time ( aPTT) ≤1.5 X ULN unless the subject is receiving anticoagulant therapy. Subjects on anticoagulant therapy must have a PT or aPTT within therapeutic range and no history of severe hemorrhage.
14. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the E7 TCR cells.. Adverse events from prior therapy must have resolved to ≤grade 1 according to CTCAE Version 5.0 or have demonstrated clinical stability for the protocol.
15. Participants must be able to understand and be willing to sign the written informed consent document.
16. Participants must agree to participate in protocol Cancer Institute of New Jersey (CINJ) 192103 (Pro2021002307) for gene therapy long term follow up and in protocol CINJ 192002 (Pro2021000281) for biospecimen collection study.

Note: Participants may have undergone minor surgical procedures with the past three weeks, as long as all toxicities have recovered to Grade 1 or less.

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from participation in this study:

1. Uncontrolled intercurrent illness such as active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
2. History of severe allergic reactions to compounds of similar chemical or biological composition to agents used in this study.
3. History of coronary revascularization or ischemic symptoms unless patient has a normal cardiac stress test.
4. Documented LVEF of less than or equal to 45% tested. The following participants will undergo cardiac evaluations:

   1. Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or
   2. Age > 50 years old
5. Participants with baseline screening pulse oxygen level of < 92% on room air will not be eligible. If the underlying cause of hypoxia improves, then they may be reevaluated.
6. Subjects with HLA-A*02:01 damaging mutation or allele loss or other molecular resistance detected by clinical or research genomic profiling will not be eligible.
7. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR T cells, breastfeeding should be discontinued if the mother is treated with E7 TCR T cells. These potential risks may also apply to other agents used in this study.
8. Participants with a systemic immunodeficiency including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune competence may be less responsive to the treatment.
9. Participants on immunosuppressive drugs including corticosteroids unless meeting criteria outlined in Section 6.1 (Prohibited Medications).
10. Participants with potentially severe autoimmune diseases such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis, autoimmune pancreatitis, or systemic lupus erythematosus are not eligible. Patients with less severe autoimmune diseases such as hypothyroidism, vitiligo, and other minor autoimmune disorders are eligible.
11. Participants with prior or concurrent malignancy whose natural history or treatment is unlikely to interfere with the safety or efficacy assessments of the investigational regimen are eligible for this trial. Examples include, but are not limited to:

    1. Carcinoma in situ
    2. Cutaneous skin cancers requiring only local excision
    3. Low grade non-muscle invasive bladder cancer
    4. Low grade prostate cancer Participants with prior or concurrent malignancy that do not meet the above criteria are excluded.
12. Subjects who received a live vaccine within 30 days prior to enrollment are not eligible.
13. Determination by the Principal Investigator that participation is not in the best interest of the research subject or may jeopardize the safety of the subject or integrity of the clinical trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response | Five years
  Objective tumor response as measured by RECIST

SECONDARY OUTCOMES:
Adverse Events | 5 years
  Adverse events as measured by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hinrichs, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Data will be made available through the publisher at the time of publication.
Access Criteria: Data will be accessible through the publisher.

REFERENCES:
- [Background] Nagarsheth NB, Norberg SM, Sinkoe AL, Adhikary S, Meyer TJ, Lack JB, Warner AC, Schweitzer C, Doran SL, Korrapati S, Stevanovic S, Trimble CL, Kanakry JA, Bagheri MH, Ferraro E, Astrow SH, Bot A, Faquin WC, Stroncek D, Gkitsas N, Highfill S, Hinrichs CS. TCR-engineered T cells targeting E7 for patients with metastatic HPV-associated epithelial cancers. Nat Med. 2021 Mar;27(3):419-425. doi: 10.1038/s41591-020-01225-1. Epub 2021 Feb 8. PMID 33558725